CLINICAL TRIAL: NCT01897662
Title: Study of the Consumption of Nutriose on Satiety, Weight Loss and Fat Mass Reducing in Overweight Subjects
Brief Title: Effect of Nutriose Supplementation on Satiety, Weight Loss and Adiposity in Overweight Subjects
Acronym: ROQ_NUTRIMETAB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nealth Sarl (Network)
Collaborators: Roquette Freres (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: ROQ_NUTRIMETAB10; 2011-A00062-39 (Registry Identifier: AFSSAPS (France))
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Overweight
Keywords: overweight; satiety; functional food; food intake; digestive tolerance
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NUTRIOSE (Experimental): Group of volunteers fed with NUTRIOSE
  Interventions: Dietary Supplement: NUTRIOSE FB06
- GLUCIDEX (Active Comparator): Group of volunteers fed with GLUCIDEX
  Interventions: Dietary Supplement: GLUCIIDEX 21

INTERVENTIONS:
Dietary Supplement: NUTRIOSE FB06 — 14g/day NUTRIOSE FB06: 7g in 250 mL orange juice twice a day
  Arms: NUTRIOSE
Dietary Supplement: GLUCIIDEX 21 — 7g/day GLUCIDEX 21 : 3.5g in 250 mL orange juice twice a day
  Arms: GLUCIDEX

SUMMARY:
NUTRIOSE is a food ingredient defined as a carbohydrate polymer of vegetable origin (wheat starch or corn) with a degree of polymerization ≥ 3 and chemically transformed. It is soluble in aqueous solution, very poorly digested in the small intestine, it mostly reaches the colon where it stimulates fermentation. AFSSA, in its opinion of July 30, 2007, considers that this ingredient is a "soluble dietary fiber." Recent work in China in overweight volunteers have shown an effect of NUTRIOSE on satiation and satiety, and demonstrate an effect on reducing weight and fat mass. By its action on satiety and reduced food intake, the NUTRIOSE be of interest in the management of overweight or obese. Among the possible mechanisms of action, are the metabolites produced by colonic fermentation of NUTRIOSE.

The goal of this biomedical research is to study the effect of a dose of 14g/day of NUTRIOSE FB06 for 12 weeks on the evolution of weight, percentage of body fat and digestive tolerance in Caucasians overweight subjects. To gather evidence to support mechanisms of action, it is proposed to measure before consumption, then every 4 weeks, the effects of NUTRIOSE FB06 on satiety and satiation and changes in colonic flora and its metabolites.

ELIGIBILITY:
Inclusion Criteria:

* healthy people
* aged between 20 and 50 years
* BMI between 27 and 29 kg/m2
* without metabolic syndrome
* no pregnant nor nursing women
* covered by Social Security
* negative serology for hepatitis B/C and HIV
* who signed the informed consent form

Exclusion Criteria:

* persons abusing drugs (laxatives, anti-diarrheal, agents acting on satiety)
* person who doesn't want to stop taking food supplements containing pre- or probiotics during time of the study
* person intolerant to gluten and / or allergic to wheat flour
* person in diet during the last 3 months
* person in vegetarian or vegan diet
* person who donated blood during the 3 months preceding the study
* Inclusion in another clinical study
* subjects receiving over 4,500 Euros in the last 12 months (including the present study)
* subjects presenting risk of non-compliance in the opinion of the recruiting doctor.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
body weight | D-7; D28; D56; D84

SECONDARY OUTCOMES:
satiety | D-7; D28; D56; D84
energy intake | D-7; D28; D56; D84
BMI | D-7; D28; D56; D84
  Body Mass Index
body fat | D-7; D28; D56; D84
  measured by DEXA
waist size | D-7; D28; D56; D84
glycemia | D-7; D28; D56; D84
insulinemia | D-7; D28; D56; D84
total cholesterol | D-7; D28; D56; D84
LDL cholesterol | D-7; D28; D56; D84
HDL cholesterol | D-7; D28; D56; D84
triglyceridemia | D-7; D28; D56; D84
HOMA | D-7; D28; D56; D84
  homeostasis model assessment (appreciates peripheral insulinoresistance and deficit in insulin secretion)
microbiota | D-7; D28; D56; D84
  measured by RT-PCR
blood pressure | D-7; D28; D56; D84
digestive tolerance | D-7; D28; D56; D84
  measured with daily questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Paul VALENSI, PU/PH, Chef de service, Principal Investigator — centre de recherche en nutrition humaine (CRNH)
Locations (1):
- CRNH, service de diabétologie-endocrinologie-nutrition hôpital Jean Verdier, Bondy, Seine-Saint-Denis, France

REFERENCES:
- [Background] Li S, Guerin-Deremaux L, Pochat M, Wils D, Reifer C, Miller LE. NUTRIOSE dietary fiber supplementation improves insulin resistance and determinants of metabolic syndrome in overweight men: a double-blind, randomized, placebo-controlled study. Appl Physiol Nutr Metab. 2010 Dec;35(6):773-82. doi: 10.1139/H10-074. PMID 21164548
- [Background] Slavin JL, Savarino V, Paredes-Diaz A, Fotopoulos G. A review of the role of soluble fiber in health with specific reference to wheat dextrin. J Int Med Res. 2009 Jan-Feb;37(1):1-17. doi: 10.1177/147323000903700101. PMID 19215668
- [Background] Guerin-Deremaux L, Li S, Pochat M, Wils D, Mubasher M, Reifer C, Miller LE. Effects of NUTRIOSE(R) dietary fiber supplementation on body weight, body composition, energy intake, and hunger in overweight men. Int J Food Sci Nutr. 2011 Sep;62(6):628-35. doi: 10.3109/09637486.2011.569492. Epub 2011 May 19. PMID 21591985
- [Background] Haarman M, Knol J. Quantitative real-time PCR assays to identify and quantify fecal Bifidobacterium species in infants receiving a prebiotic infant formula. Appl Environ Microbiol. 2005 May;71(5):2318-24. doi: 10.1128/AEM.71.5.2318-2324.2005. PMID 15870317
- [Background] Suzuki K, Simpson KA, Minnion JS, Shillito JC, Bloom SR. The role of gut hormones and the hypothalamus in appetite regulation. Endocr J. 2010;57(5):359-72. doi: 10.1507/endocrj.k10e-077. Epub 2010 Apr 14. PMID 20424341
- [Background] Ruskone-Fourmestraux A, Attar A, Chassard D, Coffin B, Bornet F, Bouhnik Y. A digestive tolerance study of maltitol after occasional and regular consumption in healthy humans. Eur J Clin Nutr. 2003 Jan;57(1):26-30. doi: 10.1038/sj.ejcn.1601516. PMID 12548293